CLINICAL TRIAL: NCT02512588
Title: A Randomized, Placebo-Controlled, Double-blind, Fixed-Dose, Multiple Cohort, Multiple Crossover, Dose-Finding Study of Oral BTD-001 in Adults With Idiopathic Hypersomnia (IH) or Narcolepsy Type 2
Brief Title: A Study of Safety and Efficacy of BTD-001 in Treatment of Patients With Idiopathic Hypersomnia (IH) or Narcolepsy Type 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Balance Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BTD-001 IH201
Record Dates: First submitted 2015-07-23; First posted 2015-07-31 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Idiopathic Hypersomnia; Narcolepsy Without Cataplexy
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BTD-001 (Experimental)
  Interventions: Drug: BTD-001
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BTD-001
  Arms: BTD-001
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind, multiple cohort, fixed-dose multiple crossover, dose-finding study of oral BTD-001 in adult patients with IH or Narcolepsy without cataplexy (Type 2).

ELIGIBILITY:
Inclusion Criteria:

* Meets ICSD-3 criteria for IH or Narcolepsy Type 2 and not undergoing pharmacologic treatment for the condition
* Usual nightly total sleep at least 6 hours as single major rest period without naps
* Epworth Sleepiness Scale of 10 or greater
* Males or females age 18 to 65 years

Exclusion Criteria:

* Any disorder causing hypersomnia other than IH or Narcolepsy Type 2
* Usual bedtime later than midnight
* Seizure disorder or history of syncope, unexplained loss of consciousness or seizure in the past 3 years
* Beck Depression Inventory score greater than 19
* Beck Anxiety Inventory score greater than 15
* Significant history of or current suicidal ideation or behavior
* BMI less than 18 kg/m2 or greater than 39 kg/m2
* Positive toxicology screen or breathalyzer test
* Clinically significant abnormal findings on safety assessments
* Any significant medical or psychiatric disease or any condition that would put the patient at risk by participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Efficacy Epworth Sleepiness Scale | After 14 days per treatment
  Epworth Sleepiness Scale

SECONDARY OUTCOMES:
Efficacy Maintenance of Wakefulness Test | After 14 days per treatment
  Maintenance of Wakefulness Test

OTHER OUTCOMES:
Pharmacokinetics (Cmax) | Selected Days 14, 35, and 56
  Pharmacokinetic parameters after multiple doses.
  -Maximum serum concentration (Cmax)
Pharmacokinetics (Tmax) | Selected Days 14, 35, and 56
  Pharmacokinetic parameters after multiple doses.
  -Time of maximum plasma concentration (Tmax)
Pharmacokinetics (T½) | Selected Days 1, 14, 31, 35, 42, and 56
  Pharmacokinetic parameters after multiple doses.
  -Elimination half life (T½)
Pharmacokinetics (AUC) | Selected Days 1, 14, 21, 35, 42, and 56
  Pharmacokinetic parameters after multiple doses.
  -Area under the concentration time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Lien, PhD, Study Director — Balance Therapeutics, Inc.
Locations (23):
- United States (23):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Stanford Medicine Sleep Center, Palo Alto, California
  - Pacific Research Network, San Diego, California
  - Empire Clinical Research, Upland, California
  - REM Sleep Medicine, Colorado Sleep Institute, Boulder, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - Emory University School of Medicine Emory Sleep Center, Atlanta, Georgia
  - NeuroTrials Research Inc, Atlanta, Georgia
  - SleepMed of Central, Macon, Georgia
  - Kentucky Research Group,, Louisville, Kentucky
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - NeuroCare Center for Sleep, Newton, Massachusetts
  - Neurological Associate, Maplewood, Minnesota
  - Clayton Sleep Institute, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Community Research Management Assoc., Cincinnati, Ohio
  - Lynn Institute, Oklahoma City, Oklahoma
  - SleepMed of South Carolina, Columbia, South Carolina
  - Future Search Trials of Neurology, Austin, Texas
  - Houston Sleep Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington